CLINICAL TRIAL: NCT06089460
Title: Longitudinal Examination of Metabolic and Behavioral Correlates of Various Protein Food Sources
Brief Title: Longitudinal Examination of Metabolic and Behavioral Correlates of Protein Sources
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-22-297-STW
Record Dates: First submitted 2023-07-28; First posted 2023-10-18 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Red Meat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beef (Experimental): Individuals will be asked to consume beef as their only source of protein and follow an individualized meal plan for 4 weeks. Thereafter, they will be instructed to continue beef consumption with any other foods desired for 4 weeks.
  Interventions: Other: Beef
- Meat analogue (Experimental): Individuals will be asked to consume a commercial meat analogue product as their only source of protein and follow an individualized meal plan for 4 weeks. Thereafter, they will be instructed to continue the meat analogue consumption with any other foods desired for 4 weeks.
  Interventions: Other: Meat analogue
- Beans/legumes (Experimental): Individuals will be asked to consume beans/legumes as their only source of protein and follow an individualized meal plan for 4 weeks. Thereafter, they will be instructed to continue the bean/legume consumption with any other foods desired for 4 weeks.
  Interventions: Other: Beans/legumes

INTERVENTIONS:
Other: Beef — Fresh, locally-sourced, grass-fed, grass-finished ground beef sufficient to meet protein needs based on body weight for 8 weeks
  Arms: Beef
Other: Meat analogue — Commercially-available and purchased meat analogue sufficient to meet protein needs based on body weight for 8 weeks
  Arms: Meat analogue
Other: Beans/legumes — Canned beans/legumes sufficient to meet protein needs based on body weight for 8 weeks
  Arms: Beans/legumes

SUMMARY:
The purpose of this three-arm, pilot, randomized controlled trial is to examine the metabolic and behavioral impacts of consuming a diet characterized by protein from red meat, a meat analogue, or beans/legumes.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age
* Willingness to consume any of the three protein sources
* Willingness to stop consumption of any pre- or pro-biotic supplements
* Willingness to follow a meal plan for four weeks

Exclusion Criteria:

* Medical condition which precludes consumption of specific foods or whole food groups

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Body weight | Baseline (week 0), T1 (week 4), T2 (week 8)
  In kilograms

SECONDARY OUTCOMES:
Fasting lipid panels (i.e., total cholesterol, HDL, LDL, VLDL, triglycerides) | Baseline (week 0), T1 (week 4), T2 (week 8)
  Total cholesterol (mg/dL), HDL (mg/dL), LDL (mg/dL), triglycerides (mg/dL)
Fasting blood glucose | Baseline (week 0), T1 (week 4), T2 (week 8)
  In mg/dL
Yale Food Addiction Scale | Baseline (week 0), T1 (week 4), T2 (week 8)
  Continuous score = 0-7 (higher = more symptoms of food addiction)
Skin carotenoids | Baseline (week 0), T1 (week 4), T2 (week 8)
Blood pressure | Baseline (week 0), T1 (week 4), T2 (week 8)
  Systolic and diastolic (mmHg)
Dietary patterns (3-day diet records) | Baseline (week 0), T1 (week 4), T2 (week 8)
Behavioral Activation Scale Reward Responsiveness | Baseline (week 0), T1 (week 4), T2 (week 8)
  Score ranges 5-20, higher scores indicate greater reward responsiveness
Ad-Libitum Ultra-Processed Food Consumption | Baseline (week 0), T1 (week 4), T2 (week 8)
  Reported in weight of food consumed, greater than or equal to 0 grams
Sensitivity to Punishment and Reward Questionnaire (Reward Questions) | Baseline (week 0), T1 (week 4), T2 (week 8)
  Score ranges 0-24, higher indicates greater sensitivity to reward

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University, Stillwater, Oklahoma, United States